CLINICAL TRIAL: NCT04871568
Title: Central Venous Stenosis Incidence After Right-sided Subclavian and Internal Jugular Vein Catheterization With a Silicone Temporary Hemodialysis Catheter
Brief Title: Central Vein Stenosis Due to Dialysis Catheter Insertion in Subclavian Compared to Jugular Vein
Acronym: CITES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Skane University Hospital (Other)
Responsible Party: Principal Investigator, Ola Borgquist, Principal Investigator, Skane University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CDC stenosis
Record Dates: First submitted 2021-04-28; First posted 2021-05-04 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Subclavian Vein Stenosis; Jugular Vein Occlusion
Keywords: Central Venous Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Right subclavian vein catheterization (Active Comparator): The temporary central dialysis catheter is placed in the right subclavian vein.
  Interventions: Procedure: Temporary central dialysis catheterization
- Right internal jugular vein catheterization (Active Comparator): The temporary central dialysis catheter is placed in the right internal jugular vein.
  Interventions: Procedure: Temporary central dialysis catheterization

INTERVENTIONS:
Procedure: Temporary central dialysis catheterization — Placement of temporary central dialysis catheter

SUMMARY:
Central vein stenosis (CVS) is a well-known complication of central venous catheterization, especially after insertion of temporary hemodialysis catheters (tHDC). Incidence and prevalence differ between studies, and exact figures are hard to tell since proper venographies seldom are performed unless the patient is symptomatic.

Most tHDC are placed in the jugular or femoral veins as catheters in the subclavian veins have been shown to result in CVS to a greater degree. However, some studies are equivocal and there are several advantages with the subclavian vein such as a lower risk for infectious and thrombotic complications, longer durability (thereby avoiding placement of a new catheter with repeated tissue trauma), increased comfort during insertion and use, less effect on blood flow if the patient moves the head, easier to mobilize.

The studies on CVS incidence originate from the 1990s when ultrasound-guided insertions were unheard of and polyurethane catheters were prevalent. The investigators believe that there is less tissue trauma when using ultrasound guidance in real-time. Furthermore, CVS is less common when silicone catheters are used instead of polyurethane catheters.

To avoid unnecessary vascular trauma and patient suffering, any pre-existing CVS should ideally be detected before cannulation attempts. A CT scan of the chest with IV contrast is preferred, but this exposes the patient to ionized radiation, is time-consuming and (although debated) may cause contrast-induced nephropathy. A brief ultrasound examination to verify central venous patency would be useful provided it is shown to have an adequate sensitivity for stenosis detection.

DETAILED DESCRIPTION:
This is a multicentric, prospective, randomized, controlled, assessor-blinded, non-inferiority trial. Patients will be enrolled in three hospitals (Lund, Malmö, Helsingborg) in southern Sweden. The trial is investigator-initiated and non-commercial. The radiologist interpreting CT venographies will be blinded to study group allocation, whereas the patient, the treating physicians and other care providers will not be blinded.

Patients will be randomized to receive a silicone tCDC either in the right subclavian vein (intervention) or in the right internal jugular vein (control). All catheterizations will be performed in a standardized manner. A questionnaire regarding the patient's experience of the catheterization procedure is handed out as soon as possible, preferably immediately after catheterization if the clinical situation permits.

Follow-up is carried out 3-6 months after the removal of the catheter to eliminate transitory thrombosis. A CT venography with a customized protocol for this study will be performed to look for CVS. An ultrasound examination of the central veins is performed and compared to the findings of the CT venography.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years of age or older).
* In need of a tCDC with an expected treatment time of at least 7 days.
* Informed consent.

Exclusion Criteria:

* Intravenous pacemaker or a PICC-line via right-sided central veins in situ.
* Known right-sided CVS.
* AV fistula on the right upper extremity.
* History of central venous vascular interventions including stents, dilatations and more (but not previous central venous catheterization).
* Central venous catheter in the right internal jugular vein or in the right subclavian vein in situ.
* Either the right jugular vein or the right subclavian vein unavailable for catheterization due to, e.g., local skin infection, thrombosis or inability to visualize the vein with ultrasound.
* Known allergy to iodinated contrast agents.
* BMI >35 kg/m2.
* No study physician available for the catheterization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Central vein stenosis | 1.5-3 months after the catheterization
  >50 percent central vein diameter reduction (stenosis) using CT venography

SECONDARY OUTCOMES:
Ultrasound-guided assessment of central vein stenosis (50 percent threshold) | 1.5-3 months after the catheterization
  Ultrasound-derived parameters indicating central vein stenosis are compared to CT venography results (with a threshold of 50 percent venous diameter reduction)
Ultrasound-guided assessment of central vein stenosis (80 percent threshold) | 1.5-3 months after the catheterization
  Ultrasound-derived parameters indicating central vein stenosis are compared to CT venography results (with a threshold of 80 percent venous diameter reduction)
Patient experience | Immediately after catheterization and 3-6 months after the catheterization
  Questionnaire regarding the patient's experience of discomfort during the catheterization procedure and when carrying the catheter
Dialysis problems | During dialysis sessions
  Blood flow rates and interruptions during dialysis are compared between the groups

CONTACTS AND LOCATIONS:
Overall Officials: Ola Borgquist, MD, PhD, Principal Investigator — Skånes universitetssjukhus; Thomas Kander, MD, PhD, Principal Investigator — Skånes universitetssjukhus
Locations (1):
- Skånes universitetssjukhus, Lund, Sweden

REFERENCES:
- [Derived] Borgquist O, Naddi L, Bozovic G, Hellberg M, Annborn M, Sjovall F, Adrian M, Hettinger E, Sjoberg P, Kander T. Central venous stenosis after subclavian versus internal jugular dialysis catheter insertion (CITES) in adults in need of a temporary central dialysis catheter: study protocol for a two-arm, parallel-group, non-inferiority randomised controlled trial. Trials. 2023 May 12;24(1):327. doi: 10.1186/s13063-023-07350-9. PMID 37173715